CLINICAL TRIAL: NCT02101320
Title: Contribution of a Hand-held Gamma Camera (TreCam) to the SNOLL(Occult Breast Lesion Localization Plus Sentinel Node Biopsy) Procedure in Breast Cancer
Brief Title: Hand-held Gamma Camera in the SNOLL Procedure
Acronym: TRECAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P120704
Record Dates: First submitted 2014-02-06; First posted 2014-04-02 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
Keywords: surgery; nuclear medicine; Lymphoscintigraphy; Gamma Camera; SNOLL; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (No Intervention): Patients with a resection of the lesions according to the procedure SNOLL without the use of TReCam.
- Group 2 (Experimental): Patients with a resection of the lesions according to the procedure SNOLL with the use of TReCam.
  Interventions: Device: TRECAM

INTERVENTIONS:
Device: TRECAM — using the camera during the surgery
  Other Names: hand held Camera
  Arms: Group 2

SUMMARY:
In France, breast cancer affects approximately 53,000 new cases per year. The investigators have to take care more and more women with subclinical lesions (nonpalpable), and it represents around 25% to 35% of the diagnosed breast cancers. The main problem of the surgical management of these lesions is the quality of preoperative identification which determines the quality of surgery and oncological and cosmetic outcomes. For this type of lesion, SNOLL (Sentinel Node and Occult Lesion Localization) procedure could be proposed. This is a radioactive labeling of the tumor site and sentinel lymph node (SLN). The investigators want to evaluate the potential benefits of using a hand held camera called TreCam in this SNOLL procedure. This camera permits to obtain nuclear imaging at the bedside and in the operating theater.

DETAILED DESCRIPTION:
Hypothesis:

The use of intraoperative TReCam improves the surgical procedure by providing relevant information during surgery to reduce the rate of further surgery for inappropriate margins.

Main Objective:

Evaluation of the contribution of TreCam in SNOLL procedure.

Main endpoint:

The rate of further surgery for inappropriate margins of the lumpectomy (less than 3mm)

Second endpoint:

Lumpectomy's characteristics, Cosmetics results Number of SLNs detected with TreCam at the different times of the procedure. Operative duration

Plan experimental :

Multicentric (3 centers) Phase II randomized non comparative study. All patients with non-palpable invasive cancer histologically proven and with ultrasound target will have SNOLL procedure.

Patients will be randomized preoperatively into two groups. Group 1: patients with a resection of the lesions according to the procedure SNOLL without the use of TReCam.

Group 2: patients with a resection of the lesions according to the procedure SNOLL with the use of TReCam.

In group 1:

* Day-1: Injection of Tc99m (Nanocis) in contact with the tumor under ultrasound guidance followed by a lymphoscintigraphy (LS): Localization and counting of the radioactive SLNs. Localization of the tumor site.
* Day 0: Before incision, exploration with the classic gamma probe (GP) for the localization of the different surgical areas (breast and axillary) is performed. Removal of SLN is achieved thanks to double detection (colorimetric and radioactive). After incision, radioactive SLN are identified by GP. At the end of the SLN procedure, the operator checks the absence of residual activity and controls with preoperative LS. In case of non detection of SLN or metastases identified during extemporaneous examination an axillary node dissection is performed. The GP is also used to guide lumpectomy and verify the absence of significant residual radioactivity after lumpectomy. Extemporaneous examination of lumpectomy specimen (size, limits of resection) is performed. Additional shaving of the cavity margins is appreciated by the surgeon.

In group 2 :

TReCam is used at different stages of SNOLL procedure:

* Day-1: A mapping with TReCam is performed after LS. (without LS results)
* Day 0: Before incision, in addition to GP, TReCam is used to define number and localization of SLN and the tumor site.

  * At the end of the usual SLN procedure, axillary area is also explored by TReCam in order to find residual SLN.
  * After lumpectomy, absence of significant residual radioactivity is checked by GP and TReCam
  * Operative duration will be reported.
  * Difficulties in data acquisition with TReCam.
  * Collection of all the histological results.
  * Outcome: Cosmetic results, decision of further surgery for inappropriate margins.

Total duration study: 13 months: Inclusion period : 12 months; Follow up : 1 month

Statistics

1. Sample size. This is a phase II 2-steps randomized non comparative study. N= 30 patients in each group. This will allow to test the potential interest of TReCAm in group 2 using an optimal II-stage design based on the number of patients without reintervention (success).

   The tested hypothesis are:

   H0: p=p0 avec p0 = 80% (poor technique) H1: p=p1>p0 avec p1 = 95% (good technique) N= 30 patients per group will be considered, method proposed by R.P. A'Hern (Stat Med 2001 :20. 859-866).

   The required power was set at 80% and the alpha risk was set at 5%.
2. Strategy analysis of data collected

   Populations studied:

   The primary analysis will focus on all randomized patients (intention to treat analysis). Given the type of patients and the evaluation time of the primary endpoint, it is unlikely that there is lost sight. However, any patient with no information available on the primary endpoint will be classified as having a reoperation.
3. Justification of statistical tests

Descriptive analysis:

All quantitative parameters will be summarized descriptively in each group of treatment modality and for each time they are collected. The analysis will include descriptive statistics for each quantitative parameter each time: average, standard deviation, minimum, maximum, median and quartiles, number of missing values. Qualitative parameters are expressed by the frequency distribution and accurate bilateral confidence intervals to 95% associated. (asymptotic estimators will not be used because of the considered effective).

ELIGIBILITY:
Inclusion Criteria :

* Patients older than 18 years
* Patients undergoing SNOLL procedure for breast non palpable invasive cancer (ultrasound image target) confirmed by biopsy before surgery
* Clinical T0N0 stage
* Before the SNOLL procedure, patients will be informed on all this procedure
* A free and informed consent must be obtained

Exclusion Criteria :

* Multifocal breast cancer, diffuse microcalcifications
* Non-palpable breast cancer without ultrasound target
* Isolated in situ cancer or invasive cancer associated with extended in situ carcinoma
* Patients who underwent neoadjuvant chemotherapy
* Palpable axillary nodes on clinical examination or with a suspicious or positive cytology
* Pregnant patient
* History of axillary surgery or mammoplasty
* Allergy to any component of the tracking technique

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Rate of further surgery for non in sano or inadequate (less than 3 mm security margins) lumpectomy piece's margins. | Between 2 and 3 weeks

SECONDARY OUTCOMES:
Size, volume and weight of the lumpectomy. | between 2 and 3 weeks
Status of resection margins | one day
  During surgery
Cosmetics results: 4 point Score | between 2 and 3 weeks
  EXCELLENT: the treated breast is almost identical to untreated breast GOOD: minor difference between the treated breast and untreated breast. FAIR: obvious difference between the treated breast and untreated breast. POOR: major aesthetic and functional sequelae in the treated breast.
Morbidity | between 2 and 3 weeks
  (hematoma, abscess...).
Volume of resection / tumor volume | between 2 and 3 weeks
  Volume of resection / tumor volume:
  (Length x width x height) specimen / (π / 6) d3.(d is the histological maximum diameter of the lesion) Length x width x height) specimen / (π / 6) d3.(d is the histological maximum diameter of the lesion
Duration of utilization of TreCam at The day before surgery and before induction of anesthesia for the location of the breast injection site and SLN. | 2 days
  The day before surgery, and at the day of surgery
Duration of utilization of TreCam at at the end of the SLN procedure for verifying the absence of radioactivity. | One Day
  Day of surgery
Duration of utilization of TreCam at each step of the procedure during the breast exploration before lumpectomy. | One day before the surgery
Duration of utilization of TreCam at at the end of lumpectomy for acquisition of images of the tumor's bed after removal of the radioactive target and for acquisition of image of the lumpectomy's specimen. | One day
  Before surgery
Difficulties in data acquisition Using a scale of 4 items : VERY EASY, EASY, DIFFICULT, IMPOSSIBLE | one day
Comparison between imaging data provided in preoperative time by TreCam and by standard LS: image's quality, location of the injection's site, location and number of SLN. | One day
  preoperative time

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre BRICOU, MD, Principal Investigator — Hôpital Jean Verdier
Locations (1):
- Service de gynécologie-Obstétrie, Bondy, France

REFERENCES:
- [Background] Barranger E, Uzan S, Pitre S, Duval MA, Charon Y. [Development of a hand-held gamma camera (POCI) in the sentinel node biopsy for breast cancer]. Pathol Biol (Paris). 2008 Jul;56(5):254-6. doi: 10.1016/j.patbio.2007.09.009. Epub 2008 Feb 21. No abstract available. French. PMID 18178328
- [Background] Medina-Franco H, Abarca-Perez L, Garcia-Alvarez MN, Ulloa-Gomez JL, Romero-Trejo C, Sepulveda-Mendez J. Radioguided occult lesion localization (ROLL) versus wire-guided lumpectomy for non-palpable breast lesions: a randomized prospective evaluation. J Surg Oncol. 2008 Feb 1;97(2):108-11. doi: 10.1002/jso.20880. PMID 18181162
- [Background] Lavoue V, Nos C, Clough KB, Baghaie F, Zerbib E, Poulet B, Lefrere Belda MA, Ducellier A, Lecuru F. Simplified technique of radioguided occult lesion localization (ROLL) plus sentinel lymph node biopsy (SNOLL) in breast carcinoma. Ann Surg Oncol. 2008 Sep;15(9):2556-61. doi: 10.1245/s10434-008-9994-y. Epub 2008 Jun 24. PMID 18574635
- [Background] Monti S, Galimberti V, Trifiro G, De Cicco C, Peradze N, Brenelli F, Fernandez-Rodriguez J, Rotmensz N, Latronico A, Berrettini A, Mauri M, Machado L, Luini A, Paganelli G. Occult breast lesion localization plus sentinel node biopsy (SNOLL): experience with 959 patients at the European Institute of Oncology. Ann Surg Oncol. 2007 Oct;14(10):2928-31. doi: 10.1245/s10434-007-9452-2. Epub 2007 Aug 1. PMID 17674108
- [Background] Kerrou K, Pitre S, Coutant C, Rouzier R, Ancel PY, Lebeaux C, Huchet V, Montravers F, Pascal O, Duval MA, Lefebvre F, Menard L, Uzan S, Charon Y, Barranger E. The usefulness of a preoperative compact imager, a hand-held gamma-camera for breast cancer sentinel node biopsy: final results of a prospective double-blind, clinical study. J Nucl Med. 2011 Sep;52(9):1346-53. doi: 10.2967/jnumed.111.090464. Epub 2011 Aug 17. PMID 21849400
- [Background] Bricou A, Duval MA, Charon Y, Barranger E. Mobile gamma cameras in breast cancer care - a review. Eur J Surg Oncol. 2013 May;39(5):409-16. doi: 10.1016/j.ejso.2013.02.008. Epub 2013 Mar 7. PMID 23465183
- [Background] The Tumor Resection Camera (TReCam), a multipixel imaging probe for radio-guided surgery.E. Netter, L. Pinot, L. Ménard, M.-A. Duval, B. Janvier, F. Lefebvre, R. Siebert, Y. Charon. Nuclear Science Symposium Conference Record (NSS/MIC), 2009 IEEE, 2573-2576